CLINICAL TRIAL: NCT02088151
Title: Selective Retinal Pigment Epithelium Laser Therapy (SRT) for Macular Disease of the Retina
Brief Title: Selective Retinal Pigment Epithelium Laser Therapy for Macular Disease of the Retina
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suitable device for laser no longer available
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003/10; 2011-MD-0006 (Other: Swissmedic)
Record Dates: First submitted 2014-03-06; First posted 2014-03-14 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Macular Edema; Central Serous Chorioretinopathy; Retinal Vein Occlusion; Age-related Macular Degeneration; Retinal Neovascularization
Keywords: selective laser therapy; retinal pigment epithelium; macular edema; diabetic retinopathy; central serous chorioretinopathy; age-related macular degeneration; retinal vein occlusion
MeSH Terms: conditions — Macular Edema; Central Serous Chorioretinopathy; Retinal Vein Occlusion; Macular Degeneration; Retinal Neovascularization; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients receive selective retinal pigment epithelium laser treatment
  Interventions: Device: Selective retinal pigment epithelium laser therapy using the R:GEN Laser System

INTERVENTIONS:
Device: Selective retinal pigment epithelium laser therapy using the R:GEN Laser System — Patients receive selective retinal pigment epithelium laser treatment using the R:GEN Laser System by Lutronic Corporation, Korea.

SUMMARY:
Laser photocoagulation of the retina targeting the outer layers is an established therapy for proliferative retinopathy and macular edema from diabetic microangiopathy or retinal vein occlusion, centrals serous retinopathy, and extrafoveal subretinal neovascular membranes. However, collateral damage occurs and scotomas can result when using conventional lasers with pulse duration of 100ms and more. This is particularly relevant for laser treatments of the macula where the main therapeutic effect results from stimulation of the retinal pigment epithelium cells and photoreceptor damage is thought to be an unnecessary side effect. Recent experimental research with new laser devices using much shorter pulse duration has shown that photoreceptor damage can be greatly reduced and the retinal pigment epithelium selectively targeted, hence the term selective retinal pigment epithelium laser therapy (SRT). Investigators hypothesize that SRT is equally effective as standard laser photocoagulation for macular disease but minimizes local visual field defects.

In this study, patients with central serous retinopathy, macular edema from diabetic microangiopathy or branch vein occlusion, and non-exudative age-related macular degeneration will be treated with SRT. Patients will be assessed 1, 3 and 6 months after treatment.

DETAILED DESCRIPTION:
Background

Laser photocoagulation of the retina targeting the outer layers is an established therapy for proliferative retinopathy and macular edema from diabetic microangiopathy or retinal vein occlusion, centrals serous retinopathy, and extrafoveal subretinal neovascular membranes. However, collateral damage occurs and scotomas can result when using conventional lasers with pulse duration of 100ms and more. This is particularly relevant for laser treatments of the macula where the main therapeutic effect results from stimulation of the retinal pigment epithelium cells and photoreceptor damage is thought to be an unnecessary side effect. Recent experimental research with new laser devices using much shorter pulse duration has shown that photoreceptor damage can be greatly reduced and the retinal pigment epithelium selectively targeted, hence the term selective retinal pigment epithelium laser therapy (SRT). In age-related macular degeneration, regression of drusen has been observed after laser treatment with convention laser or SRT. Investigators hypothesize that SRT is equally effective as standard laser photocoagulation for macular disease but minimizes local visual field defects.

Objective

To assess the efficacy of SRT in patients with central serous retinopathy, macular edema from diabetic microangiopathy or branch vein occlusion, and non-exudative age-related macular degeneration. Up to five patients with proliferative diabetic retinopathy can optionally be treated with SRT too.

Methods

At baseline and during follow-up patients will receive a full ophthalmic examination including optical coherence tomography, fundus autofluorescence imaging, fluorescein angiography (FA), and visual acuity testing. SRT (R:GEN Laser System by Lutronic Corporation, Korea) will be delivered under topical anesthesia. For titration of energy spots will first be applied outside the major arcades. Immediately thereafter FA will be performed for extrapolation of the laser dose, since the treatment is sub-threshold and laser spots will not be visible biomicroscopically. The patient will then be treated at the discretion of the ophthalmologist with up to 500 laser burns. One hour after the laser treatment FA will be repeated to confirm the treatment effect. Patients will be assessed 1, 3 and 6 months after treatment. Pulse duration can be chosen between 200ns and 2μs. The maximum pulse energy will be 1mJ. 1-30 pulses will be applied for every laser burn at a frequency of 100Hz.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Written informed consent
* Willingness to attend follow-up visits
* Central serous chorioretinopathy affecting visual acuity
* Macular edema from branch retinal vein occlusion
* Macular edema from diabetic microangiopathy
* Age-related macular degeneration with confluent soft drusen
* Age-related macular degeneration with geographic atrophy

Exclusion Criteria

* Macular ischemia
* Retinal hemorrhage impeding retinal laser treatment
* Subretinal neovascular membrane
* Vitreous hemorrhage
* Allergy to fluorescein
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-06; Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Visual Acuity according to ETDRS protocol | 6 months

SECONDARY OUTCOMES:
Retinal thickness measured by optical coherence tomography | 6 months
Leakage of fluorescein in fluorescein angiography | 6 months
Area of absent fundus autofluorescence | 6 months
  Measured via fundus autofluorescence imaging

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolf, Study Chair — Department of Ophthalmology, Bern University Hospital; Andreas Ebneter, Principal Investigator — Department of Ophthalmology, Bern University Hospital
Locations (1):
- Department of Ophthalmology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Roider J, Michaud NA, Flotte TJ, Birngruber R. Response of the retinal pigment epithelium to selective photocoagulation. Arch Ophthalmol. 1992 Dec;110(12):1786-92. doi: 10.1001/archopht.1992.01080240126045. PMID 1463423
- [Background] Roider J, Hillenkamp F, Flotte T, Birngruber R. Microphotocoagulation: selective effects of repetitive short laser pulses. Proc Natl Acad Sci U S A. 1993 Sep 15;90(18):8643-7. doi: 10.1073/pnas.90.18.8643. PMID 8378341
- [Background] Roider J, Lindemann C, el-Hifnawi el-S, Laqua H, Birngruber R. Therapeutic range of repetitive nanosecond laser exposures in selective RPE photocoagulation. Graefes Arch Clin Exp Ophthalmol. 1998 Mar;236(3):213-9. doi: 10.1007/s004170050067. PMID 9541826
- [Background] Roider J, Brinkmann R, Wirbelauer C, Birngruber R, Laqua H. Variability of RPE reaction in two cases after selective RPE laser effects in prophylactic treatment of drusen. Graefes Arch Clin Exp Ophthalmol. 1999 Jan;237(1):45-50. doi: 10.1007/s004170050193. PMID 9951641
- [Background] Roider J, Brinkmann R, Wirbelauer C, Laqua H, Birngruber R. Subthreshold (retinal pigment epithelium) photocoagulation in macular diseases: a pilot study. Br J Ophthalmol. 2000 Jan;84(1):40-7. doi: 10.1136/bjo.84.1.40. PMID 10611098